CLINICAL TRIAL: NCT01810952
Title: The Management of Glucocorticoid-Induced Hyperglycemia in Hospitalized Patients
Acronym: GIH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Glenn R. Cunningham, Professor of Medicine and Molecular & Cellular Biology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-27172
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Hyperglycemia; Diabetes Mellitus
Keywords: glucocorticoids; hyperglycemia; diabetes mellitus
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus | interventions — Insulin Glargine; Insulin Lispro; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glargine/Lispro Insulin Arm (Experimental): Drug: Glargine insulin was administered per above.
  Drug: Lispro insulin 0.2 unit/kg/day was administered per above. A "coverage" dose of 0.1 unit/kg/day of lispro for each 10 mg of prednisone or its equivalent was divided between 3 meals. The maximum starting "coverage" dose was 0.4 units/kg per day.
  The prandial dose of lispro was increased by 10% if the pre-lunch, pre-dinner, or bedtime SG was between 141-200 mg/dL, and by 20% if the pre-lunch, pre-dinner or bedtime SG is >200 mg/dL. The prandial dose of lispro was decreased by 10% if the pre-lunch, pre-dinner, or bedtime SG is between 70-89 mg/dL, and by 20% if the pre-lunch, pre-dinner or bedtime SG was less than 70 mg/dL.
  Drug: prednisone or equivalent dose was determined by severity of exacerbation and clinician's judgement.
  Interventions: Drug: Glargine insulin; Drug: Lispro insulin
- Glargine/Lispro/NPH Insulin Arm (Experimental): Drugs Glargine and Lispro insulin included similar starting doses of glargine and lispro.
  Drug: A "coverage" dose of NPH insulin 0.1 unit/kg/day for each 10 mg of prednisone or its equivalent was given twice daily with the administration of the glucocorticoid. Maximum starting "coverage" dose was 0.4 units/kg per day. NPH dose was increased by 10% if the pre-lunch, pre-dinner, or bedtime SG is between 141-200 mg/dL, and by 20% if the pre-lunch, pre-dinner or bedtime SG was greater than 200 mg/dL. It was decreased by 10% if the pre-lunch, pre-dinner, or bedtime SG was between 70-89 mg/dL, and by 20% if the pre-lunch, pre-dinner or bedtime SG was less than 70 mg/dL.
  Drug: the dose of prednisone or equivalent glucocorticoid was determined by severity of exacerbation and clinician's judgement.
  Interventions: Drug: Glargine insulin; Drug: Lispro insulin; Drug: NPH Insulin

INTERVENTIONS:
Drug: Glargine insulin — In both protocols glargine dose was increased by 10% if the FSG value was 141-200 mg/dL and by 20% if the FSG value was more than 200 mg/dL, and decreased by 10% if the FSG was 70-89 mg/dL and by 20% if the FSG was less than 70 mg/dL.
Drug: Lispro insulin — In both protocols lispro insulin was given to cover meals. Additional lispro insulin was Lispro insulin was administered before meals to cover the prednisone or glucocorticoid equivalent in the Glargine/Lispro Insulin Arm.
Drug: NPH Insulin — NPH insulin was given once or twice a day to cover the prednisone or glucocorticoid equivalent in the Glargine/Lispro/NPH Insulin Arm
  Arms: Glargine/Lispro/NPH Insulin Arm

SUMMARY:
The investigators hypothesize that includes patient weight and glucocorticoid dose can be used to safely initiate insulin treatment in diabetic/hyperglycemic patients who are to be treated with pharmacological doses of glucocorticoids.

DETAILED DESCRIPTION:
The target fasting serum glucose (FSG) and pre-meal SG was 90-140 mg/dL, and the random SG was less than 180 mg/dL, taking into consideration the ADA/AACE target glucose levels in non-ICU patients (15).

The Glargine/Lispro Protocol included 0.2 unit/kg/day as insulin glargine once daily if the dose was between 40-80 units, or twice daily if the dose was less than 40 or more than 80 units; plus 0.2 unit/kg/day as lispro divided between three meals for all insulin-naïve patients. A "coverage" dose of 0.1 unit/kg/day of lispro for each 10 mg of prednisone or its equivalent was divided between 3 meals. The maximum starting "coverage" dose was 0.4 units/kg per day.

The prandial dose of lispro was increased by 10% if the pre-lunch, pre-dinner, or bedtime SG was between 141-200 mg/dL, and by 20% if the pre-lunch, pre-dinner or bedtime SG is >200 mg/dL. The prandial dose of lispro was decreased by 10% if the pre-lunch, pre-dinner, or bedtime SG is between 70-89 mg/dL, and by 20% if the pre-lunch, pre-dinner or bedtime SG was less than 70 mg/dL.

The Glargine/Lispro/NPH Protocol included 0.2 unit/kg/day as insulin glargine as per G/L; plus 0.2 unit/kg/day as lispro divided between three meals for all the insulin-naïve patients. A "coverage" dose of 0.1 unit/kg/day of Neutral Protamine Hagedorn (NPH) for each 10 mg of prednisone or its equivalent was given twice daily with the administration of the glucocorticoid. The maximum starting "coverage" dose was 0.4 units/kg per day.

The NPH dose was increased by 10% if the pre-lunch, pre-dinner, or bedtime SG is between 141-200 mg/dL, and by 20% if the pre-lunch, pre-dinner or bedtime SG was greater than 200 mg/dL. The NPH dose was decreased by 10% if the pre-lunch, pre-dinner, or bedtime SG was between 70-89 mg/dL, and by 20% if the pre-lunch, pre-dinner or bedtime SG was less than 70 mg/dL.

In both protocols glargine dose was increased by 10% if the fasting glucose value is 141-200 mg/dL and by 20% if the fasting glucose value was more than 200 mg/dL, and decreased by 10% if the FSG was 70-89 mg/dL and by 20% if the FSG was less than 70 mg/dL.

If the patient had an outpatient regimen which includes a total daily dose of insulin (TDI) that exceeded 0.4 unit/kg/day, then the same TDI was continued with 50% given as glargine once daily if the dose was between 40-80 units, or twice daily if the dose was less than 40 or more than 80 units; and 50% given as lispro divided between three meals. The patient was still randomly assigned to either one of the two protocols as described previously.

If the patient were on a TDI less than 0.4 unit/kg/day in addition to oral antidiabetic medications as an outpatient, then all the oral antidiabetic medications were discontinued and the patient was started on 0.5 unit/kg/day divided as 50% glargine given once daily if the dose was between 40-80 units, or twice daily if the dose was less than 40 or more than 80 units; and 50% lispro divided between three meals. The patient was randomly assigned to either one of the two protocols based upon even and odd hospital numbers.

ELIGIBILITY:
Inclusion Criteria:

* Admission for Chronic Obstructive Pulmonary Disease (COPD) exacerbation.
* Treatment with pharmacological doses of glucocorticoids (GCs) ≥10 mg of prednisone or its equivalent if they are not on maintenance dose of GCs in the outpatient settings.
* Treatment with pharmacological doses of GCs ≥10 mg of prednisone or its equivalent above their maintenance dose of GCs in the outpatient settings.
* Have either a previous diagnosis of diabetes mellitus which has been treated with diet or medications, hemoglobin A1c ≥6.5%, or confirmed inpatient hyperglycemia defined as a fasting laboratory glucose or finger stick reading ≥126 mg/dL or random glucose reading ≥200 mg/dL on two or more determinations.

Exclusion Criteria:

Unwilling to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn R Cunningham, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- St. Luke's Episcopal Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clore JN, Thurby-Hay L. Glucocorticoid-induced hyperglycemia. Endocr Pract. 2009 Jul-Aug;15(5):469-74. doi: 10.4158/EP08331.RAR. PMID 19454391
- [Background] Moghissi ES, Korytkowski MT, DiNardo M, Einhorn D, Hellman R, Hirsch IB, Inzucchi SE, Ismail-Beigi F, Kirkman MS, Umpierrez GE; American Association of Clinical Endocrinologists; American Diabetes Association. American Association of Clinical Endocrinologists and American Diabetes Association consensus statement on inpatient glycemic control. Diabetes Care. 2009 Jun;32(6):1119-31. doi: 10.2337/dc09-9029. Epub 2009 May 8. No abstract available. PMID 19429873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified from admission listing of patients and admitting diagnoses. Admitting physician was contacted to determine eligibility and if s/he were agreeable to our approaching patient regarding the study. Protocol was explained to patient. If s/he agreed to participate, they were asked to sign an informed consent.
Groups:
- Glargine/Lispro Insulin: The Glargine/Lispro Arm included 0.2 unit/kg/day as insulin glargine daily if the dose was between 40-80 units, or twice daily if the dose was less than 40 or more than 80 units; plus 0.2 unit/kg/day as lispro divided between three meals for all insulin-naïve patients. A "coverage" dose of 0.1 unit/kg/day of lispro for each 10 mg of prednisone or its equivalent was divided between 3 meals. The maximum starting "coverage" dose was 0.4 units/kg per day.
  Glargine/Lispro insulin: In both protocols glargine dose was increased by 10% if the fasting glucose value was 141-200 mg/dL and by 20% if the fasting glucose value was more than 200 mg/dL, and decreased by 10% if the fasting FSG was 70-89 mg/dL and by 20% if the fasting FSG was less than 70 mg/dL.
- Glargine/Lispro/NPH Insulin: The basal and prandial doses of glargine and lispro insulin were similar to those in the Glargine/Lispro Arm. A "coverage" dose of 0.1 unit/kg/day of NPH for each 10 mg of prednisone or its equivalent was given twice daily with the administration of the glucocorticoid. The maximum starting "coverage" dose was 0.4 units/kg per day.
Period: Overall Study
Arm/Group | Glargine/Lispro Insulin | Glargine/Lispro/NPH Insulin
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Glargine/Lispro Insulin Arm: The Glargine/Lispro Arm included 0.2 unit/kg/day as insulin glargine daily if the dose was between 40-80 units, or twice daily if the dose was less than 40 or more than 80 units; plus 0.2 unit/kg/day as lispro divided between three meals for all insulin-naïve patients. A "coverage" dose of 0.1 unit/kg/day of lispro for each 10 mg of prednisone or its equivalent was divided between 3 meals. The maximum starting "coverage" dose was 0.4 units/kg per day.
  Glargine/Lispro insulin: In both protocols glargine dose was increased by 10% if the fasting glucose value was 141-200 mg/dL and by 20% if the fasting glucose value was more than 200 mg/dL, and decreased by 10% if the fasting FSG was 70-89 mg/dL and by 20% if the fasting FSG was less than 70 mg/dL.
- Glargine/Lispro/NPH Insulin Arm: The basal and prandial doses of glargine and lispro insulin were similar to those in the Glargine/Lispro Arm. A "coverage" dose of 0.1 unit/kg/day of NPH for each 10 mg of prednisone or its equivalent was given twice daily with the administration of the glucocorticoid. The maximum starting "coverage" dose was 0.4 units/kg per day.
- Total: Total of all reporting groups
Arm/Group | Glargine/Lispro Insulin Arm | Glargine/Lispro/NPH Insulin Arm | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 6 | 19
  >=65 years | 7 | 11 | 18
Age, Continuous [Mean (Standard Deviation); unit: years]
  Baseline Participants | 60.8 (12.9) | 67.1 (14.3) | 63.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Glucose Levels on Days 1-5 After the Initiation of the Treatment Protocol.
Description: Most patients had 4 and all patients had at least 2 readings each day. Average daily glucose values were determined for each participant, then averaged for each Arm."
Time Frame: 1-5 days
Population: We used t-tests to compare values between the protocols on each day..
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Glargine/Lispro Insulin Arm: The G/L Arm will include 0.2 unit/kg/day as insulin glargine daily if the dose is between 40-80 units, or twice daily if the dose is less than 40 or more than 80 units; plus 0.2 unit/kg/day as lispro divided between three meals for all insulin-naïve patients. A "coverage" dose of 0.1 unit/kg/day of lispro for each 10 mg of prednisone or its equivalent will be divided between 3 meals. The maximum starting "coverage" dose will be 0.4 units/kg per day.
  Glargine/Lispro insulin: In both protocols glargine dose will be increased by 10% if the fasting glucose value is 141-200 mg/dL and by 20% if the fasting glucose value is more than 200 mg/dL, and decreased by 10% if the fasting FSG is 70-89 mg/dL and by 20% if the fasting FSG is less than 70 mg/dL.
- Glargine/Lispro/NPH Insulin Arm: Basal and meal coverage for G/L/N Arm is similar to that in the GL Arm. A "coverage" dose of 0.1 unit/kg/day of NPH for each 10 mg of prednisone or its equivalent will be given twice daily with the administration of the glucocorticoid. The maximum starting "coverage" dose will be 0.4 units/kg per day.
  Glargine/Lispro/NPH insulin: The G/L/N Protocol will include 0.2 unit/kg/day as insulin glargine daily if the dose is between 40-80 units, or twice daily if the dose is less than 40 or more than 80 units; plus 0.2 unit/kg/day as lispro divided between three meals for all the insulin-naïve patients. A "coverage" dose of 0.1 unit/kg/day of NPH for each 10 mg of prednisone or its equivalent will be given twice daily with the administration of the glucocorticoid. The maximum starting "coverage" dose will be 0.4 units/kg per day.
Arm/Group | Glargine/Lispro Insulin Arm | Glargine/Lispro/NPH Insulin Arm
Number analyzed (Participants) | 20 | 17
mg/dL
  Day 1 (n=20, 17) | 181.8 (40.9) | 173.7 (51.2)
  Day 2 (n=20, 17) | 160.5 (45.5) | 148.4 (36.7)
  Day 3 (n=20, 17) | 155.1 (51.8) | 140.8 (35.2)
  Day 4 (n=14, 12) | 159.5 (40.5) | 133.4 (34.0)
  Day 5 (n=10, 7) | 151.7 (45.5) | 132.0 (33.5)
Statistical Analysis 1: Comparison: Glargine/Lispro Insulin Arm vs Glargine/Lispro/NPH Insulin Arm; Test type: Superiority or Other; p = 0.35, t-test, 2 sided — This is the p-value for Day 5

2. Secondary Outcome: Percent of Participants With Average Glucose >70 and <180 mg/dL
Description: Percent of Participants with Average Daily Glucose >70 and <180 mg/dL
Time Frame: Last Full Day of Protocol for Participant (up to Day 5)
Measure: Number; unit: percentage of participants
Groups:
- Glargine/Lispro Insulin Arm; Glargine/Lispro/NPH Insulin Arm: Last Full Day of Protocol
Arm/Group | Glargine/Lispro Insulin Arm | Glargine/Lispro/NPH Insulin Arm
Number analyzed (Participants) | 20 | 17
percentage of participants | 90 | 94
Statistical Analysis 1: Comparison: Glargine/Lispro Insulin Arm vs Glargine/Lispro/NPH Insulin Arm; Test type: Superiority or Other; p = 0.65, Chi-squared

3. Secondary Outcome: Daily Insulin Dose/Kg Body Weight
Description: Total daily dose of insulin required based on weight and glucocorticoid dosage to achieve average daily finger stick glucose (FSG) levels of 90-140 mg/dL
Time Frame: 1-5 days
Measure: Mean (Standard Deviation); unit: units of insulin/Kg body weight
Groups:
- Glargine/Lispro Insulin Arm; Glargine/Lispro/NPH Insulin Arm: Insulin (units)/kg body weight
Arm/Group | Glargine/Lispro Insulin Arm | Glargine/Lispro/NPH Insulin Arm
Number analyzed (Participants) | 20 | 17
units of insulin/Kg body weight
  Day 1 (n=20, 17) | 0.89 (0.25) | 0.80 (0.17)
  Day 2 (n=20, 17) | 0.91 (0.28) | 0.82 (0.18)
  Day 3 (n=20, 17) | 0.96 (0.35) | 0.77 (0.24)
  Day 4 (n=14, 12) | 1.01 (0.50) | 0.75 (0.16)
  Day 5 (n=10, 7) | 1.12 (0.70) | 0.65 (0.21)
Statistical Analysis 1: Comparison: Glargine/Lispro Insulin Arm vs Glargine/Lispro/NPH Insulin Arm; Daily values for each protocol were compared using t-tests; Test type: Superiority or Other; p = 0.06, t-test, 2 sided — Comparison of the 5 day averages resulted in a p-value of 0.06

4. Secondary Outcome: Glucose Values <70 mg/dL.
Description: # participants with glucose values <70 mg/dL
Time Frame: 1-5 days
Measure: Number; unit: participants
Arm/Group | Glargine/Lispro Insulin Arm | Glargine/Lispro/NPH Insulin Arm
Number analyzed (Participants) | 20 | 17
participants
  # with glucose values <70 mg/dL | 5 | 4
  # with glucose values <60 mg/dL | 4 | 2
  # with glucose <50 | 1 | 0
Statistical Analysis 1: Comparison: Glargine/Lispro Insulin Arm vs Glargine/Lispro/NPH Insulin Arm; Test type: Superiority or Other; p = 0.795, Chi-squared — Comparison of the number of participants in each group with glucose value <70 mg/dL resulted in p-value 0.795; difference in binomial proportions

5. Post Hoc Outcome: Percent of Glucose Determinations >180 mg/dL
Time Frame: 1-5 days
Measure: Number; unit: Percent of glucose values
Arm/Group | Glargine/Lispro Insulin Arm | Glargine/Lispro/NPH Insulin Arm
Number analyzed (Participants) | 20 | 17
Percent of glucose values | 31.0 | 24.6
Statistical Analysis 1: Comparison: Glargine/Lispro Insulin Arm vs Glargine/Lispro/NPH Insulin Arm; Values in each group were compared by Chi squared; Test type: Superiority or Other; p = 0.055, Chi-squared — Comparison between groups of percent of glucose values >180 mg/dL

ADVERSE EVENTS:
Groups:
- Glargine/Lispro Insulin Arm: The G/L Arm received 0.2 unit/kg/day as insulin glargine daily if the dose was between 40-80 units, or twice daily if the dose was less than 40 or more than 80 units; plus 0.2 unit/kg/day as lispro divided between three meals for all insulin-naïve patients. A "coverage" dose of 0.1 unit/kg/day of lispro for each 10 mg of prednisone or its equivalent was divided between 3 meals. The maximum starting "coverage" dose was 0.4 units/kg per day.
  Glargine/Lispro insulin: In both protocols glargine dose was increased by 10% if the fasting glucose value was 141-200 mg/dL and by 20% if the fasting glucose value was more than 200 mg/dL, and decreased by 10% if the fasting FSG was 70-89 mg/dL and by 20% if the fasting FSG was less than 70 mg/dL.
- Glargine/Lispro/NPH Insulin Arm: The basal and prandial doses of glargine and lispro were similar to those in the G/L/N Protocol. A "coverage" dose of 0.1 unit/kg/day of NPH for each 10 mg of prednisone or its equivalent was given twice daily with the administration of the glucocorticoid. The maximum starting "coverage" dose was 0.4 units/kg per day.
Arm/Group | Glargine/Lispro Insulin Arm | Glargine/Lispro/NPH Insulin Arm
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/17
Other Adverse Events (participants affected / at risk) | 0/20 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine/Lispro Insulin Arm (N=20) | Glargine/Lispro/NPH Insulin Arm (N=17)
Glucose value <50 mg/dL. (Endocrine disorders) | 1 (1) | 0 (0) — This occurred when she received lispro insulin and then failed to eat.

LIMITATIONS AND CAVEATS:
The number of participants is limited, and some were discharged in less than 5 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No